CLINICAL TRIAL: NCT02575898
Title: Feasibility of a Creative Writing Intervention in an Advanced Cancer Population: A Single Arm, Consecutive Cohort Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Dartmouth-Hitchcock Medical Center (Other)
Responsible Party: Principal Investigator, Maxwell. T. Vergo, Staff Physician, Palliative Care, Dartmouth-Hitchcock Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: D15113
Record Dates: First submitted 2015-10-08; First posted 2015-10-15 (Estimated); Last update posted 2018-11-19 (Actual); Status verified 2018-11

CONDITIONS: Primary Malignant Neoplasm of Lung; Primary Malignant Neoplasm of Gastrointestinal Tract
MeSH Terms: conditions — Lung Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- One (Other): Creative writing and questionnaires interventions:
  First Session, Second Session, Third through Sixth Sessions
  Interventions: Other: First Session; Other: Second Session; Behavioral: Third through Sixth Sessions

INTERVENTIONS:
Other: First Session — Creative Practice and Positive Re-enforcement
Other: Second Session — Disease Related
Behavioral: Third through Sixth Sessions — Life Review and Legacy

SUMMARY:
To assess the feasibility of a creative writing intervention in an advanced cancer population. Given it is a relatively simple intervention delivered by a non-clinician, the investigators are interested in better understanding its pattern of effect on patient psychological adjustment. The investigators aim to assess its feasibility in this study in order to inform a future larger study that will utilize a control arm.

DETAILED DESCRIPTION:
Participants will be recruited within 3 months of presenting with a new GI or lung primary, non-curable malignancy. After consent, the participants will meet with the staff writer, who is already part of the creative arts program, to determine the methods, themes and modalities of creative writing to pursue. These choices will be revisited each session, as patients move from one theme to another, and some patients may consistently choose a given modality such as letters, while others will choose variety.

Participants will meet with the staff writer one-on-one by scheduled appointment in the outpatient or inpatient setting at a minimum of once per month throughout a 6 month time period after enrollment. This appointment is preferred to be in person, but due to the rural setting may be conducted by telephone if needed. There will not be a protocol regarding the length of and number of visits during the 6 month study period, but these quantities will be recorded to use for analysis of effectiveness of the intervention.

Writing modality choices will include private thoughts and feelings in a journal, poetry, letters to oneself or loved ones and narrative writing about significant life events. All interventions will focus on a written product for the participant to have and potentially share with caregivers if they desire.

Every 3 months patients will be asked to complete the following series of questionnaires: ECOG PS, PGAC3, HADS4, DT5, CSE6, CD-RISC-107, PTGI-SF8, FACIT-Sp-Ex9, ESAS11 and PA10.

Patients will be followed for 9 months after enrollment or until death (whichever is soonest). If a patient decides to discontinue the creative writing intervention before 6 months, the reason will be recorded and they will continue in the study for 9 months or until death completing the questionnaires.

Anyone completing the first intervention with the creative writer will be evaluable for the feasibility outcome. If the investigators see 50% of patients completing 3 months of the creative writing intervention then this would indicate the intervention should be examined in a larger pilot study. In addition, the investigators will carefully record accrual rate with associated reasons for declining and number of patients able to complete the full planned intervention with the creative writing. In planning for a larger pilot study next and given the survey burden is high in this study, the investigators will plan to use a subset analysis in order to see which factors were significantly affected by the creative arts intervention

ELIGIBILITY:
Inclusion Criteria:

1. Participant must plan to receive follow up care at Dartmouth-Hitchcock.
2. Participant must have a lung or GI primary cancer diagnosed in the last 3 months.
3. Participant must have non-curable cancer as judged by the primary oncologist.
4. Participant must be comfortable conversing in English (reading and writing in English is not required).
5. Participant must be cognitively intact as judged by their responsible clinician.
6. Participant must have access to a working telephone and be willing and available to participate by this modality as needed.
7. Participants may be on anti-depressants and/or anxiolytics as long as the dosing has remained stable over the preceding 2 weeks.

Exclusion Criteria:

1. Participant is expected to die in 6 months or less as judged by the responsible clinician.
2. Participant must not have already worked with the staff writer at Dartmouth Hitchcock prior to enrollment in this study.
3. Participant with an activated durable power of attorney for health care or cognitive impairment that interferes with ability to understand prognosis as determined by the primary oncologist.
4. Participant must not have uncontrolled physical symptoms.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2016-01-14 (Actual); Primary Completion 2018-07-12 (Actual); Study Completion 2018-09-04 (Actual)

PRIMARY OUTCOMES:
Feasibility of a creative writing intervention in an advanced cancer population | 29 months
  Anyone completing the first intervention with the creative writer will be evaluable for the feasibility outcome. If the investigators see 50% of patients completing 3 months of the creative writing intervention then this would indicate the intervention should be examined in a larger pilot study.

CONTACTS AND LOCATIONS:
Overall Officials: Max Vergo, MD, Principal Investigator — Dartmouth-Hitchcock Medical Center
Locations (1):
- Dartmouth-Hitchcock Medical Center, Lebanon, New Hampshire, United States

REFERENCES:
- [Background] Temel JS, Greer JA, Muzikansky A, Gallagher ER, Admane S, Jackson VA, Dahlin CM, Blinderman CD, Jacobsen J, Pirl WF, Billings JA, Lynch TJ. Early palliative care for patients with metastatic non-small-cell lung cancer. N Engl J Med. 2010 Aug 19;363(8):733-42. doi: 10.1056/NEJMoa1000678. PMID 20818875
- [Background] Temel JS, Greer JA, Admane S, Gallagher ER, Jackson VA, Lynch TJ, Lennes IT, Dahlin CM, Pirl WF. Longitudinal perceptions of prognosis and goals of therapy in patients with metastatic non-small-cell lung cancer: results of a randomized study of early palliative care. J Clin Oncol. 2011 Jun 10;29(17):2319-26. doi: 10.1200/JCO.2010.32.4459. Epub 2011 May 9. PMID 21555700
- [Background] Greer JA, Pirl WF, Jackson VA, Muzikansky A, Lennes IT, Heist RS, Gallagher ER, Temel JS. Effect of early palliative care on chemotherapy use and end-of-life care in patients with metastatic non-small-cell lung cancer. J Clin Oncol. 2012 Feb 1;30(4):394-400. doi: 10.1200/JCO.2011.35.7996. Epub 2011 Dec 27. PMID 22203758
- [Background] Bakitas MA, Tosteson TD, Li Z, Lyons KD, Hull JG, Li Z, Dionne-Odom JN, Frost J, Dragnev KH, Hegel MT, Azuero A, Ahles TA. Early Versus Delayed Initiation of Concurrent Palliative Oncology Care: Patient Outcomes in the ENABLE III Randomized Controlled Trial. J Clin Oncol. 2015 May 1;33(13):1438-45. doi: 10.1200/JCO.2014.58.6362. Epub 2015 Mar 23. PMID 25800768
- [Background] Bakitas M, Lyons KD, Hegel MT, Balan S, Brokaw FC, Seville J, Hull JG, Li Z, Tosteson TD, Byock IR, Ahles TA. Effects of a palliative care intervention on clinical outcomes in patients with advanced cancer: the Project ENABLE II randomized controlled trial. JAMA. 2009 Aug 19;302(7):741-9. doi: 10.1001/jama.2009.1198. PMID 19690306
- [Background] Dionne-Odom JN, Azuero A, Lyons KD, Hull JG, Tosteson T, Li Z, Li Z, Frost J, Dragnev KH, Akyar I, Hegel MT, Bakitas MA. Benefits of Early Versus Delayed Palliative Care to Informal Family Caregivers of Patients With Advanced Cancer: Outcomes From the ENABLE III Randomized Controlled Trial. J Clin Oncol. 2015 May 1;33(13):1446-52. doi: 10.1200/JCO.2014.58.7824. Epub 2015 Mar 23. PMID 25800762
- [Background] Bohlmeijer E, Smit F, Cuijpers P. Effects of reminiscence and life review on late-life depression: a meta-analysis. Int J Geriatr Psychiatry. 2003 Dec;18(12):1088-94. doi: 10.1002/gps.1018. PMID 14677140
- [Background] Chochinov HM, Hack T, Hassard T, Kristjanson LJ, McClement S, Harlos M. Dignity therapy: a novel psychotherapeutic intervention for patients near the end of life. J Clin Oncol. 2005 Aug 20;23(24):5520-5. doi: 10.1200/JCO.2005.08.391. PMID 16110012
- [Background] Ando M, Tsuda A, Morita T. Life review interviews on the spiritual well-being of terminally ill cancer patients. Support Care Cancer. 2007 Feb;15(2):225-31. doi: 10.1007/s00520-006-0121-y. Epub 2006 Sep 12. PMID 16967303
- [Background] Steinhauser KE, Alexander SC, Byock IR, George LK, Olsen MK, Tulsky JA. Do preparation and life completion discussions improve functioning and quality of life in seriously ill patients? Pilot randomized control trial. J Palliat Med. 2008 Nov;11(9):1234-40. doi: 10.1089/jpm.2008.0078. PMID 19021487
- [Background] Crogan NL, Evans BC, Bendel R. Storytelling intervention for patients with cancer: part 2--pilot testing. Oncol Nurs Forum. 2008 Mar;35(2):265-72. doi: 10.1188/08.ONF.265-272. PMID 18321839
- [Background] Chochinov HM, Kristjanson LJ, Breitbart W, McClement S, Hack TF, Hassard T, Harlos M. Effect of dignity therapy on distress and end-of-life experience in terminally ill patients: a randomised controlled trial. Lancet Oncol. 2011 Aug;12(8):753-62. doi: 10.1016/S1470-2045(11)70153-X. Epub 2011 Jul 6. PMID 21741309
- [Background] Puetz TW, Morley CA, Herring MP. Effects of creative arts therapies on psychological symptoms and quality of life in patients with cancer. JAMA Intern Med. 2013 Jun 10;173(11):960-9. doi: 10.1001/jamainternmed.2013.836. PMID 23699646
- [Background] Korte J, Bohlmeijer ET, Cappeliez P, Smit F, Westerhof GJ. Life review therapy for older adults with moderate depressive symptomatology: a pragmatic randomized controlled trial. Psychol Med. 2012 Jun;42(6):1163-73. doi: 10.1017/S0033291711002042. PMID 21995889
- [Background] Juliao M, Oliveira F, Nunes B, Vaz Carneiro A, Barbosa A. Efficacy of dignity therapy on depression and anxiety in Portuguese terminally ill patients: a phase II randomized controlled trial. J Palliat Med. 2014 Jun;17(6):688-95. doi: 10.1089/jpm.2013.0567. Epub 2014 Apr 15. PMID 24735024
- [Background] Tegner I, Fox J, Philipp R, et al. Evaluating the use of poetry to improve well-being and emotional resilience in cancer patients. J Poetry Ther 2009; 22: 121-131.